CLINICAL TRIAL: NCT05617326
Title: Screening for Abdominal Aortic Aneurysms in the General Practice by Ultraportable Ultrasound: Cluster Randomized Controlled Prospective Multicenter Study in Two Parallel Groups 1:1 in Open-label
Brief Title: Screening for Abdominal Aortic Aneurysms in the General Practice by Ultraportable Ultrasound
Acronym: DACEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HPD_2022_8
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- screening by a GP (Experimental): Each patient in this group will have a screening for AAA performed by a trained general practitioner
  Interventions: Other: AAA screening by a GP
- screening by a radiologist (conventional) (Other): Each patient in this group will have AAA screening performed by a radiologist
  Interventions: Other: AAA screening by a radiologist

INTERVENTIONS:
Other: AAA screening by a GP — The GPs included in the experimental group will be trained in AAA screening with an ultra-portable ultrasound machine and will keep an ultrasound machine available (Butterfly iQ+ model). Their patients will be able to be screened by the GP in the office or at home. In case of positive screening, the GP will be able to refer the patients to the radiologist for diagnostic confirmation..
  Arms: screening by a GP
Other: AAA screening by a radiologist — General practitioners in the control group will refer their patients to the radiologist for AAA screening.
  Arms: screening by a radiologist (conventional)

SUMMARY:
Abdominal aortic aneurysm (AAA) is a localized dilatation of a segment of the aorta artery in its abdominal portion. It affects 1.7% of men aged 65 years and older. In the high-risk population (male smokers aged 65-75 years), its prevalence is estimated to be between 2.8 and 9%. Mortality of ruptured AAAs is high (80% of deaths before hospitalization or perioperatively), whereas mortality of scheduled procedures for unruptured AAAs is less than 5%. AAA screening has been shown to significantly reduce the specific mortality rate in the medium and long term. The French National Authority for Health (HAS) recommends targeted screening for AAA by ultrasound at the radiologist. The target population is male smokers or former smokers aged 65 to 75 years, as well as all persons aged 50 to 75 years with a family history of AAA. Despite recommendations, the rate of access to targeted screening appears low. Ultrasound screening for AAA is a rapid, noninvasive, and reproducible test. It relies primarily on the measurement of the maximum diameter of the abdominal aorta in cross-section. It has been demonstrated that the learning of the ultrasound screening procedure for AAA is very fast and that the performance of non-radiologists trained in this procedure alone is similar to that of radiologists.

In addition, new ultra-portable ultrasound devices, inexpensive and with validated performances have appeared on the market in the last few years, making it possible to equip general practitioners (GPs). We propose a simplified care pathway for AAA screening, by equipping GPs with an ultra-portable ultrasound scanner and by training them to perform the screening procedure, which will be performed in the office or at the patient's home, during a usual consultation of general medicine. Our hypothesis is that this new organization will allow better access to screening for the target population, at a lower cost, compared to the current screening method recommended by the HAS (referral of the patient to the radiologist).

ELIGIBILITY:
Inclusion Criteria:

* Male
* In the absence of a family history of AAA: Patient aged 65 to 75 years, chronic current or past smoker, active smoker (defined as having smoked at least one cigarette per day) or former smoker (defined as having quit smoking less than 20 years ago, regardless of the number of cigarettes smoked).
* If there is a family history of AAA: Patient between 50 and 75 years of age
* Express consent to participate in the study
* Affiliated or beneficiary of a social security plan

Exclusion Criteria:

* Patient with a legal protection measure
* Patient with previous AAA screening less than 5 years old
* Patient unable to understand the study / give informed consent (cognitive impairment, communication impairment)

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
AAA screening performed at 1 year | 1 year
  Percentage of included patients (eligible for AAA screening) who actually received AAA screening ultrasound within 1 year of the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Picard, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (5):
- France (5):
  - Cabinet IPSO Brotteaux, Lyon
  - Cabinet IPSO Saint Martin, Paris
  - Cabinet IPSO Nation, Paris
  - Cabinet IPSO Italie, Paris
  - Cabinet IPSO Ourcq, Paris